CLINICAL TRIAL: NCT05336201
Title: The Cognitive-Remediation of Executive and Adaptive Deficits in Youth (C-READY) Intervention: a Randomized Controlled Trial for Adolescents with Sickle Cell Disease to Prepare for Transition of Care
Brief Title: Cognitive Remediation Intervention to Prepare for Transition of Care
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Donna Murdaugh, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 300003655
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease; Cognitive Impairment; Adolescent Behavior; Self Efficacy; Health-Related Behavior; Coping Skills
MeSH Terms: conditions — Anemia, Sickle Cell; Cognitive Dysfunction; Adolescent Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-READY (Cognitive-Remediation of Executive and Adaptive Deficits in Youth) (Experimental): Self-management and goal-setting cognitive remediation
  Interventions: Behavioral: CREADY (Cognitive-Remediation of Executive and Adaptive Deficits in Youth)
- Wait-List Control Group (Other): Will receive the same C-READY intervention after a 4-week wait period
  Interventions: Behavioral: CREADY (Cognitive-Remediation of Executive and Adaptive Deficits in Youth)

INTERVENTIONS:
Behavioral: CREADY (Cognitive-Remediation of Executive and Adaptive Deficits in Youth) — Manualized cognitive remediation intervention that includes 1) skills-based remediation (metacognitive training), 2) parent training, and 3) cognitive behavioral approaches. Intervention targets self-management and goal-setting skill building to promote independence in activities necessary for transition of care.

SUMMARY:
Randomized Controlled Trial (RTC) testing the efficacy of a telehealth adaptation of the Cognitive-Remediation of Executive and Adaptive Deficits in Youth (C-READY) intervention to prepare adolescents with sickle cell disease for transition of care.

DETAILED DESCRIPTION:
Cognitive impairment is a pervasive debilitating feature of sickle cell disease (SCD), with over 50% of children demonstrating early neurodevelopmental delays, ultimately influencing ability for adolescents with SCD to engage in effective decision-making needed for successful transition into adulthood. The negative effect of cognitive impairment on transition to adult self-care is further compounded by health-related disparities and poor social determinants of health. Transition to self-care among youth with SCD may be facilitated by cognitive remediation. One potential avenue to disseminate cognitive-based interventions to disadvantaged neighborhoods is through telehealth administration. This study will examine the efficacy of C-READY on adaptive and self-management skills in youth with SCD, where there is a critical need to enhance self-efficacy/self-care skills for successful transition into adulthood. Additionally, this study overcomes the barriers of transportation that preclude vulnerable patient populations from returning to the clinic for in-person interventions by offering the intervention in their homes via telehealth. C-READY is a manualized, individualized intervention delivered over the course of 4 weeks in 8, 60 minute one-on-one telehealth sessions between the youth and trained therapist. Caregiver involvement and accountability is promoted by weekly phone sessions in between the 8 primary sessions. The emphasis C-READY is on promotion of independence with adaptive skills necessary for transition of care to adult healthcare, such as managing medications, pain management, sleep hygiene, and/or daily health-related routines; the objective is to identify and focus on goals that best promote those skills. Thus, we will conduct a two-arm, wait-listed randomized control trial among 120 patients with SCD (ages 10-18 years), 60 participants per group; half randomized to the intervention arm, and half to the waitlist arm. The primary outcome is transition readiness skills, with secondary outcome measures of cognitive abilities and neuroimaging metrics. We hypothesize that youth with SCD who participate in C-READY will show improvement in transition readiness skills and show greater improvement in cognitive performance. We also hypothesize that participation in C-READY will improve functional brain connectivity and increase compensatory neural mechanisms. In sum, this study will be the first step in developing highly accessible and scalable evidence-based intervention to improve transition of care, enhance self-care, and ultimately improve overall quality of life in youth with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD (all genotypes)
* Active follow-up at Children's of Alabama Hospital
* Ages 10-18
* English-speaking

Exclusion Criteria:

* History of seizures or overt stroke
* History of Intellectual Disability or Autism Spectrum Disorder
* Inability to participate in the MRI scan, such as metal implants, neurostimulators, claustrophobia
* Currently on psychotropic medications

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Transition Readiness | 4-weeks
  Questionnaire assessing how knowledgeable the youth is about their health condition and the skills necessary for self-management and self-advocacy
Transition Readiness | 4-months post-intervention
  Questionnaire assessing how knowledgeable the youth is about their health condition and the skills necessary for self-management and self-advocacy

SECONDARY OUTCOMES:
Cognitive Assessment | 4-weeks
  A global cognitive deficit score will be calculated that assesses intellectual functioning, working memory, processing speed, attention, language, and executive functioning. The global cognitive deficit score is calculated as an average of test scores and normalized to a scale of 0-5, with 0 indicating normal functioning and 5 indicating severe deficits.
Cognitive Assessment | 4-months post-intervention
  A global cognitive deficit score will be calculated that assesses intellectual functioning, working memory, processing speed, attention, language, and executive functioning. The global cognitive deficit score is calculated as an average of test scores and normalized to a scale of 0-5, with 0 indicating normal functioning and 5 indicating severe deficits.
Neuroimaging | 4-weeks
  Brain scan (MRI) of structural and functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Sharing of the data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. We will also make our results available to other scientists interested in understanding cognitive outcomes in youth with sickle cell disease, and to avoid unintentional duplication of research. We also hope that the results of this study will lead to future collaboration to further develop approaches to improve transition of care outcomes in adolescents and youth adults with sickle cell disease. Our plan includes presentation at national and international meetings and publications in peer-reviewed medical journals. All publications of these data will contain a statement of data sharing so that other researchers will know of its availability.